CLINICAL TRIAL: NCT05677529
Title: Prodromal and Overt Parkinson's Disease Epidemiological Study in Brazil
Acronym: PROBE-PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Artur Francisco Schuh, MD, PhD, Hospital de Clinicas de Porto Alegre
Other Study IDs: MJFF-020850
Record Dates: First submitted 2022-08-10; First posted 2023-01-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Parkinsonism
Keywords: Parkinson's disease; Prodromal symptoms; Neurodegenerative disorder; REM Sleep Behavior Disorder; Primary parkinsonism; Epidemiology; Health Disparity, Minority and Vulnerable Populations; Risk Factors; Parkinsonian Disorders; Prevalence
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Prodromal Symptoms; Neurodegenerative Diseases; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Hair and blood samples will be collected from a subsample of volunteers screened positive and negative after presential neurological consultation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson's Disease (PD) affects people universally, including all ethnic and socioeconomic groups, as a highly prevalent neurodegenerative disorder. However, there are several additional challenges for people living with PD in developing countries, especially those with low socioeconomic status. There is limited access to neurological care in Brazil due to an uneven distribution of neurologists and neurological facilities, which is more critical in the poorest regions. In addition, people in these vulnerable communities are more exposed to environmental pollution, including pesticides and metals used in agriculture and mining, respectively. Therefore, reliable data on the prevalence and incidence of PD in Brazil are essential to understand the proportion of this limited access to care for patients with PD, its burden in the region, and the potential role of environmental and lifestyle risk factors in PD. Unfortunately, the literature describes few epidemiological data on PD in Latin America, including Brazil, with an evident need for more information in their regions remarkably different. The investigators will carry out a population-based study in four municipalities in Brazil (Veranópolis-RS, Belém-PA, Jacobina-BA and Candangolândia-DF), comprising distinct communities in terms of ethnic groups, education levels, and environmental and lifestyle exposures, to portray the differences in Brazilian society. The present study will screen all people living in these regions aged 60 and over for parkinsonian symptoms and REM sleep behavior disorder (RBD). At least one neurologist will examine those selected to determine the diagnosis of PD or related disorders. The study also will evaluate a random sample of those individuals with a negative screen. Each participant selected after the screening will undergo clinical assessments and interview with the addition of a comprehensive questionnaire on clinical and sociodemographic data, prodromal symptoms, as well as lifestyle and environmental exposures, including occupational use and non-occupational use of pesticides and metals. An equal sample of blood and hair will be collected from individuals with PD and controls. The study will determine the prevalence of PD and related disorders in these distinct communities. An exploratory analysis also will be performed to determine the association between PD and each variable investigated.

DETAILED DESCRIPTION:
Detailed Description:

This project proposes to evaluate the prevalence of PD and other parkinsonian syndromes in four regions of Brazil. Additionally, the incidence of PD and conversion of premotor symptoms into parkinsonian syndromes will be investigated in a 5-year cohort in a population-based sample in the southern region country. The investigators will also perform an exploratory analysis to assess the effect of environmental and lifestyle risk factors on PD.

Primary Purpose:

To determine the prevalence of Parkinson's disease and other Parkinson's syndromes in population-based samples of people aged 60 and over in the cities of Veranópolis (RS), Belém (PA), Jacobina (BA), and the administrative region of Candangolândia (DF).

Secondary Objective:

For all four regions studied:

To determine the overall prevalence and age- and sex-adjusted prevalence of Parkinson's disease; To determine the prevalence of other forms of parkinsonism (atypical, drug and vascular parkinsonism); To determine the prevalence of pre-motor symptoms of Parkinson's disease (REM sleep behavior disorder (RBD), constipation, hyposmia, subtle voice changes, depression in a sample of elderly individuals) To assess the association between Parkinson's disease and exposure to environmental factors: caffeine, tobacco, alcohol, pesticides, herbicides and other environmental toxicants; To evaluate the association between Parkinson's disease and biochemical and molecular biomarkers in peripheral fluids. The biological markers will be uric acid, iron, ferritin, transferrin and heavy metals;

Data Analysis Methodology:

The investigators will follow the STROBE statement for cross-sectional studies for data analysis and reporting of results for the study of prevalence and risk factors (Vandenbroucke et al. 2014). Data collection will be recorded in spreadsheets and digitally captured by REDCap tools (Harris et al. 2009) hosted at Hospital de Clínicas de Porto Alegre. For PD and other parkinsonian disorders, the aim will be to estimate: 1) crude prevalence, 2) age-specific prevalence, 3) gender-specific prevalence, and 4) age-adjusted prevalence rate.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older;
* Permanent residence in Veranópolis, Candangolândia, Jacobina or Islands of Belém.

Exclusion Criteria:

* Under 60 years of age
* Not have permanent residence in Veranópolis, Candangolândia, Jacobina or Islands of Belém.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population-based observational study to identify parkinsonian syndromes in four Brazilian cities: (1) Veranópolis, located in southern Brazil, with 25,936 inhabitants and an HDI of 0.773; (2) the insular portion of Belém (Ilha do Mosqueiro - Sucurijuquara and Furo das Marinhas Districts, Ilha do Outeiro - District of Fama, Combu and Cotijuba Islands), in the Amazon, Northern Brazil, with 15,469 inhabitants and an HDI of 0.573; (3) Candangolândia, in the Center-West of Brazil, with 16,196 inhabitants and an HDI of 0.852; and (4) Jacobina, in the Northeast of Brazil, with 80,635 inhabitants and an HDI of 0,649. All are small to medium-sized communities from different Brazilian regions, with different ethnic and socioeconomic compositions, which capture part of the country's diversity.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of parkinsonian syndrome and Parkinson's disease | The estimated time to apply Tanner and REM sleep behavior disorder (RBD) questionnaire for each study participant will be 10-15 minutes. Clinical assessment, questionnaire response, and blood and hair collection will take approximately 1.5 hours.
  All people aged 60 and over will be screened for parkinsonian symptoms by the Tanner questionnaire (composed of 10 yes or no questions about motor signs). In addition, a questionnaire (RBD1Q) will be applied, consisting of one question that assesses REM sleep behavior disorder (RBD). The selected participants will undergo clinical assessments and interview with the aid of a comprehensive questionnaire on clinical and sociodemographic data, prodromal symptoms, as well as environmental and lifestyle exposures, including occupational and non-occupational use of pesticides and metals. A neurologist dedicated to Movement Disorders will diagnose parkinsonian syndrome based on the presence of bradykinesia plus rigidity or rest tremor and PD diagnosis based on the MDS Diagnostic Criteria. We will calculate for each region the (1) crude prevalence, (2) age-specific prevalence, (3) gender-specific prevalence, and (4) age-adjusted prevalence rate.

SECONDARY OUTCOMES:
Prevalence of secondary parkinsonisms, atypical parkinsonian syndromes, subtle parkinsonism of uncertain significance, suspected REM sleep behavior disorder | The neurological assessment and application of the MDS-UPDRS for each study participant is estimated to take 10 to 15 minutes. Clinical and neurological assessment, questionnaire response and blood and hair collection will take approximately 1.5 hours.
  Participants selected in the screening will be evaluated by a neurologist dedicated to Movement Disorders with the aim of identifying any neurological condition other than parkinsonian syndrome, from a neurological assessment and application of the MDS-UPDRS.

OTHER OUTCOMES:
MDS - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | The estimated time to apply the MDS-UPDRS will be 30 minutes.
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale. It is a rating tool designed to assess the course of Parkinson's disease progression in patients. Each rating ranges from 0 to 4. The total score is between 0 and 108, the sum of 27 observation scores.
REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ) | The estimated time to apply the REM Sleep Behavior Disorder Screening Questionnaire will be 30 minutes.
  A single-question screen for Idiopathic rapid eye movement (REM) Sleep Behavior Disorder (RBD).
Montreal Cognitive Assessment (MoCA) | The estimated time to apply the Montreal Cognitive Assessment (MoCA) will be 10 minutes.
  The MoCA is a cognitive screening test designed to assist Health Professionals in the detection of mild cognitive impairment. Scores range from 0-30.
Beck Depression Inventory (BDI-II) | The estimated time to apply the Beck Depression Inventory (BDI-II) will be 10 minutes.
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression).
Environmental exposure questionnaire | The estimated time to apply the Environmental exposure questionnaire will be 30 minutes.
  The questionnaire assess the following exposures: specific medications, tobacco, alcohol, soda, black tea, source of drinking water, trauma, occupation, heavy metals, pesticides and fish intake.
Sociodemographic questionnaire | The estimated time to apply the sociodemographic questionnaire will be 30 minutes.
  Clinical and Sociodemographic Assessment Questionnaire assess sociodemographic information, which includes age, gender, family history, smoking, exposure to pesticides, comorbidities, medications in use, history of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Artur F Schuh-Schumacher, Dr., Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (4):
- Brazil (4):
  - Hospital Geral Roberto Santos, Salvador, Estado de Bahia
  - Hospital Sírio Libanês, Brasília, Federal District
  - Instituto de Ciências da Saúde, Belém, Pará
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barbosa MT, Caramelli P, Maia DP, Cunningham MC, Guerra HL, Lima-Costa MF, Cardoso F. Parkinsonism and Parkinson's disease in the elderly: a community-based survey in Brazil (the Bambui study). Mov Disord. 2006 Jun;21(6):800-8. doi: 10.1002/mds.20806. PMID 16482566
- [Background] Ball N, Teo WP, Chandra S, Chapman J. Parkinson's Disease and the Environment. Front Neurol. 2019 Mar 19;10:218. doi: 10.3389/fneur.2019.00218. eCollection 2019. PMID 30941085
- [Background] Berg D, Postuma RB, Adler CH, Bloem BR, Chan P, Dubois B, Gasser T, Goetz CG, Halliday G, Joseph L, Lang AE, Liepelt-Scarfone I, Litvan I, Marek K, Obeso J, Oertel W, Olanow CW, Poewe W, Stern M, Deuschl G. MDS research criteria for prodromal Parkinson's disease. Mov Disord. 2015 Oct;30(12):1600-11. doi: 10.1002/mds.26431. PMID 26474317
- [Background] Beck AT, Steer RA, Carbin MG. Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical Psychology Review. 1º de janeiro de 1988;8(1):77-100.
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468
- [Background] Bovolenta TM, de Azevedo Silva SM, Arb Saba R, Borges V, Ferraz HB, Felicio AC. Systematic Review and Critical Analysis of Cost Studies Associated with Parkinson's Disease. Parkinsons Dis. 2017;2017:3410946. doi: 10.1155/2017/3410946. Epub 2017 Mar 5. PMID 28357150
- [Background] Caldas ED, Jardim AN. Exposure to toxic chemicals in the diet: is the Brazilian population at risk? J Expo Sci Environ Epidemiol. 2012 Jan-Feb;22(1):1-15. doi: 10.1038/jes.2011.35. Epub 2011 Oct 12. PMID 21989502
- [Background] Consensus statement on the definition of orthostatic hypotension, pure autonomic failure, and multiple system atrophy. J Neurol Sci. 1996 Dec;144(1-2):218-9. No abstract available. PMID 8994128
- [Background] Elbaz A, Carcaillon L, Kab S, Moisan F. Epidemiology of Parkinson's disease. Rev Neurol (Paris). 2016 Jan;172(1):14-26. doi: 10.1016/j.neurol.2015.09.012. Epub 2015 Dec 21. PMID 26718594
- [Background] GBD 2016 Parkinson's Disease Collaborators. Global, regional, and national burden of Parkinson's disease, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):939-953. doi: 10.1016/S1474-4422(18)30295-3. Epub 2018 Oct 1. PMID 30287051
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Guigoz Y. The Mini Nutritional Assessment (MNA) review of the literature--What does it tell us? J Nutr Health Aging. 2006 Nov-Dec;10(6):466-85; discussion 485-7. PMID 17183419
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Heinzel S, Berg D, Gasser T, Chen H, Yao C, Postuma RB; MDS Task Force on the Definition of Parkinson's Disease. Update of the MDS research criteria for prodromal Parkinson's disease. Mov Disord. 2019 Oct;34(10):1464-1470. doi: 10.1002/mds.27802. Epub 2019 Aug 14. PMID 31412427
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Khan S, Nabi G, Naeem M, Ali L, Silburn PA, Mellick GD. A door-to-door survey to estimate the prevalence of Parkinsonism in Pakistan. Neuropsychiatr Dis Treat. 2016 Jun 21;12:1499-506. doi: 10.2147/NDT.S86329. eCollection 2016. PMID 27382292
- [Background] Khedr EM, Fawi G, Abbas MA, Mohammed TA, El-Fetoh NA, Attar GA, Zaki AF. Prevalence of Parkinsonism and Parkinson's disease in Qena governorate/Egypt: a cross-sectional community-based survey. Neurol Res. 2015 Jul;37(7):607-18. doi: 10.1179/1743132815Y.0000000020. Epub 2015 Mar 23. PMID 25796953
- [Background] Lahrmann H, Cortelli P, Hilz M, Mathias CJ, Struhal W, Tassinari M. EFNS guidelines on the diagnosis and management of orthostatic hypotension. Eur J Neurol. 2006 Sep;13(9):930-6. doi: 10.1111/j.1468-1331.2006.01512.x. PMID 16930356
- [Background] Lima CT, Freire AC, Silva AP, Teixeira RM, Farrell M, Prince M. Concurrent and construct validity of the audit in an urban brazilian sample. Alcohol Alcohol. 2005 Nov-Dec;40(6):584-9. doi: 10.1093/alcalc/agh202. Epub 2005 Sep 5. PMID 16143704
- [Background] Machado TH, Fichman HC, Santos EL, Carvalho VA, Fialho PP, Koenig AM, Fernandes CS, Lourenco RA, Paradela EMP, Caramelli P. Normative data for healthy elderly on the phonemic verbal fluency task - FAS. Dement Neuropsychol. 2009 Jan-Mar;3(1):55-60. doi: 10.1590/S1980-57642009DN30100011. PMID 29213611
- [Background] Melcon MO, Anderson DW, Vergara RH, Rocca WA. Prevalence of Parkinson's disease in Junin, Buenos Aires Province, Argentina. Mov Disord. 1997 Mar;12(2):197-205. doi: 10.1002/mds.870120210. PMID 9087978
- [Background] Montalvo Herdoíza Juan Paúl, Albear Toala Lisbeth Estefanía, Intriago Mercado Elba Rosa, Moreira-Vera Diana Victoria, Montalvo Perero Paola Susana. Prevalencia De La Enfermedad De Parkinson: Estudio Puerta-Puerta En La Provincia De Manabí-Ecuador. Rev Ecuat Neurol [Internet]. 2017 Abr [citado 2022 Jul 27] ; 26( 1 ): 23-26. Disponible en: http://scielo.senescyt.gob.ec/scielo.php?script=sci_arttext&pid=S2631-25812017000300023&lng=es.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Nicoletti A, Sofia V, Bartoloni A, Bartalesi F, Gamboa Barahon H, Giuffrida S, Reggio A. Prevalence of Parkinson's disease: a door-to-door survey in rural Bolivia. Parkinsonism Relat Disord. 2003 Oct;10(1):19-21. doi: 10.1016/s1353-8020(03)00066-x. PMID 14499202
- [Background] Opasso PR, Barreto SD, Ortiz KZ. Phonemic verbal fluency task in adults with high-level literacy. Einstein (Sao Paulo). 2016 Jul-Sep;14(3):398-402. doi: 10.1590/S1679-45082016AO3629. PMID 27759830
- [Background] Pena-Pereira MA, Sobreira-Neto MA, Sobreira E, Chagas MHN, Oliveira DS, Rodrigues GR, Souza CP, Eckeli AL, Fernandes RMF, Tumas V. Validation of the Brazilian Portuguese version of the Rapid Eye Movement Sleep Behavior Disorder Screening Questionnaire (RBDSQ-BR). Arq Neuropsiquiatr. 2020 Oct;78(10):629-637. doi: 10.1590/0004-282X20200125. Epub 2020 Oct 28. PMID 33146233
- [Background] Postuma RB, Arnulf I, Hogl B, Iranzo A, Miyamoto T, Dauvilliers Y, Oertel W, Ju YE, Puligheddu M, Jennum P, Pelletier A, Wolfson C, Leu-Semenescu S, Frauscher B, Miyamoto M, Cochen De Cock V, Unger MM, Stiasny-Kolster K, Fantini ML, Montplaisir JY. A single-question screen for rapid eye movement sleep behavior disorder: a multicenter validation study. Mov Disord. 2012 Jun;27(7):913-6. doi: 10.1002/mds.25037. Epub 2012 May 30. PMID 22729987
- [Background] Potashkin J, Huang X, Becker C, Chen H, Foltynie T, Marras C. Understanding the links between cardiovascular disease and Parkinson's disease. Mov Disord. 2020 Jan;35(1):55-74. doi: 10.1002/mds.27836. Epub 2019 Sep 4. PMID 31483535
- [Background] Pringsheim T, Jette N, Frolkis A, Steeves TD. The prevalence of Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2014 Nov;29(13):1583-90. doi: 10.1002/mds.25945. Epub 2014 Jun 28. PMID 24976103
- [Background] Dorsey ER, Bloem BR. The Parkinson Pandemic-A Call to Action. JAMA Neurol. 2018 Jan 1;75(1):9-10. doi: 10.1001/jamaneurol.2017.3299. No abstract available. PMID 29131880
- [Background] Rocha GH, Lini RS, Barbosa F Jr, Batista BL, de Oliveira Souza VC, Nerilo SB, Bando E, Mossini SA, Nishiyama P. Exposure to heavy metals due to pesticide use by vineyard farmers. Int Arch Occup Environ Health. 2015 Oct;88(7):875-80. doi: 10.1007/s00420-014-1010-1. Epub 2014 Dec 31. PMID 25549625
- [Background] Santos, Walberto Silva dos, Valdiney Veloso Gouveia, Darlene Pinho Fernandes, Sarah Stella Bomfim de Souza, and Alex Sandro de Moura Grangeiro. 2012. "Alcohol Use Disorder Identification Test (AUDIT): explorando seus parâmetros psicométricos." Jornal brasileiro de psiquiatria 61 (3): 117-23.
- [Background] Schneider Medeiros M, P Reddy S, P Socal M, Schumacher-Schuh AF, Mello Rieder CR. Occupational pesticide exposure and the risk of death in patients with Parkinson's disease: an observational study in southern Brazil. Environ Health. 2020 Jun 17;19(1):68. doi: 10.1186/s12940-020-00624-8. PMID 32552814
- [Background] Spielberger, Charles Donald. 1999. STAXI-2: State-Trait Anger Expression Inventory-2 : Professional Manual. Psychological Assessment Resources.
- [Background] Tangamornsuksan W, Lohitnavy O, Sruamsiri R, Chaiyakunapruk N, Norman Scholfield C, Reisfeld B, Lohitnavy M. Paraquat exposure and Parkinson's disease: A systematic review and meta-analysis. Arch Environ Occup Health. 2019;74(5):225-238. doi: 10.1080/19338244.2018.1492894. Epub 2018 Nov 25. PMID 30474499
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. Int J Surg. 2014 Dec;12(12):1500-24. doi: 10.1016/j.ijsu.2014.07.014. Epub 2014 Jul 18. PMID 25046751
- [Background] Zini LB, Gutterres M. Chemical contaminants in Brazilian drinking water: a systematic review. J Water Health. 2021 Jun;19(3):351-369. doi: 10.2166/wh.2021.264. PMID 34152292
- [Background] Power, Mick, WHOQOL-OLD Group, Kathryn Quinn, and Silke Schmidt. 2015. "World Health Organization Quality of Life-Old Module." PsycTESTS Dataset.
- See also: Câncer, Instituto Nacional D. O. 2015. "Posicionamento Do INCA Acerca Dos Agrotóxicos." INCA Brasília-DF — https://www.inca.gov.br/sites/ufu.sti.inca.local/files//media/document//posicionamento-do-inca-sobre-os-agrotoxicos-06-abr-15.pdf
- See also: Carmo, Marina Araujo Trajano do, Luiz Claudio Meirelles, and Ariany Oliveira Santos Nicolich. 2018. Análise do Programa de Análise de Resíduos de Agrotóxicos em Alimentos (PARA) no período de 2010 a 2016 no Brasil. ABRASCO. — https://www.arca.fiocruz.br/bitstream/icict/38462/2/Marina_Araujo_Trajano_do_Carmo.pdf
- See also: Carneiro, Fernando Ferreira, and Others. 2015. Dossiê ABRASCO: Um Alerta Sobre Os Impactos Dos Agrotóxicos Na Saúde. EPSJV/Expressão Popular. — https://www.arca.fiocruz.br/bitstream/icict/26221/2/Livro%20EPSJV%20013036.pdf